CLINICAL TRIAL: NCT02891343
Title: Effect of Hypoxia on Cognitive Assessment and Cerebral Activity in Healthy Volunteers WP1 P002 PHARMACOG
Brief Title: Effect of Hypoxia on Cognitive Assessment and Cerebral Activity in Healthy Volunteers
Acronym: Hypoxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013_44; 2014-A00513-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Alteration of Cognitive Function; Hypoxia
Keywords: Cognitive Function; Hypoxia; Neurophysiological Function; Effect of Alzheimer Disease symptomatic drugs; Healthy Subjects
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Other: 2-hour period of hypoxia

INTERVENTIONS:
Other: 2-hour period of hypoxia — During this period, the FiO2 will be set on 21% (normoxia condition). A filter will be put between the mask and the tubes connecting it to the machine generating hypoxia (equipment reference = Altitrainer NP190). On that filter a gas analyser will monitor the FiO2 and a capnography monitor (Capnostream 20, ORIDION) will also be installed.

SUMMARY:
The early assessment of new symptomatic drugs for Alzheimer disease remains difficult because of the lack of predictive end-point. The use of a battery including different parameters could improve this early development. In healthy volunteers, to test the reverse effect of symptomatic drugs, it is necessary to induce transient and reversible cognitive impairment and cerebral activity changes by a challenge test. In this context, a transient hypoxia could be relevant.

ELIGIBILITY:
Inclusion Criteria:

* Good health on the basis of the medical interview, physical examination and standard biology parameters.
* Right-Handed
* Non-smoker
* No cardiac nor pulmonary pathologies
* No use of chronic treatment or psychotropic drugs or substances
* BMI inferior to 25 Kg/m2
* French speaker and able to understand the test instructions
* Informed consent form signed

Exclusion Criteria:

1. Subject with history or current brain disease (severe brain trauma, transient ischemic attack, stroke, epilepsy, cerebral tumor…) or retinal pathologies (including familial DMLA)
2. Subject with history of Acute Mountain Sickness, High Altitude Cerebral Edema or High Altitude Pulmonary Edema
3. Subject with other major medical or surgical history including coronaropathy and pulmonary arterial hypertension
4. Subject with current chronic disease
5. Subject with vascular or metabolic risk factor
6. Subject with history of or current mental disease or addiction (MINI)
7. Subject with significant abnormality on biology
8. Subject with significant abnormality on ECG
9. Subject with significant abnormality on MRI
10. Subject with significant abnormality of electrical activities on EEG
11. Subject with family history of young onset dementia
12. Subject with family history of cardiac or pulmonary pathologies
13. Subject with family history of chronic or severe neurological or mental disease (first degree relatives)
14. Subject with claustrophobia or contraindication to MRI
15. Subject under guardianship
16. Subject not covered by Social Security
17. Subject participating in another clinical trial
18. Subject with anxiety (STAI-Trait Score T> 51) or neuroticism personality (EPI Score N ≥13)
19. Subject bearded or refusing to shave

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
the mean of response latency to the Rapid Visual Information Processing (RVIP) test of the CANTAB battery | Between baseline (normoxic period) and Day 0 (hypoxia session )

SECONDARY OUTCOMES:
The number of adverse events occuring during the period of hypoxia | at the baseline and after the hypoxia session (day0)

CONTACTS AND LOCATIONS:
Overall Officials: Régis Bordet, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Centre d'Investigation Clinique, CHRU, Lille
  - Centre d'investigation Clinique, Marseille

IPD SHARING:
Plan to Share IPD: No